CLINICAL TRIAL: NCT05417490
Title: Research Into Factors Determining Participation in Two Interventions Modifying the Care Pathways of Patients With Heart Failure in Eastern Occitanie: PRADO-IC and Telemedicine
Brief Title: Research Into Factors Determining Participation in 2 Interventions Modifying the Care Pathways of Patients With Heart Failure: PRADO and Telemedicine
Acronym: PARTI-PARC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0018
Record Dates: First submitted 2022-06-02; First posted 2022-06-14 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure
Keywords: heart failure; transitional care; PRADO; remote monitoring
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group with PRADO: All patients seen in hospital and for whom the doctor will choose whether or not to offer one of the 2 solutions, alone or in combination, will be considered as included in the study, and their non-objection will be collected.
  Subsequently, patients will benefit from follow-up for 6 months: V0 inclusion visit- V1 telephone contact at 1 month only for patients participating in one of the 2 programs and V2 consultation at 6 months. The 0 and 6M (6 months) visits are part of the usual follow-up of patients hospitalized for heart failure.
  Administration of questionnaires:
  * Girerd's questionnaire : The objective is to measure the medication compliance of patients during treatment
  * SSQ6 (Social Support Questionnaire 6) : which measures two dimensions of social support (satisfaction and availability). SSQ6 is an abbreviated form of SSQ (Social Support Questionnaire). A high SSQ score indicates more optimism about life than a low score.
  Interventions: Other: PRADO-IC
- Group with PRADO + remote monitoring: All patients seen in hospital and for whom the doctor will choose whether or not to offer one of the 2 solutions, alone or in combination, will be considered as included in the study, and their non-objection will be collected.
  Subsequently, patients will benefit from follow-up for 6 months: V0 inclusion visit- V1 telephone contact at 1 month optional only for patients participating in one of the 2 programs and V2 consultation at 6 months. The 0 and 6M visits are part of the usual follow-up of patients hospitalized for heart failure.
  Administration of questionnaires:
  * Girerd's questionnaire
  * SUTAQ (Service User Technology Acceptability Questionnaire) : only for patients with remote monitoring.
  the questionnaire has 22 items, measured on a Likert scale from 1 to 6, reflecting respectively more or less agreement with the statements of the items. The questionnaire has 5 subscales, each containing between 3 and 9 items.
  * SSQ6
  Interventions: Other: PRADO-IC; Device: Remote monitoring
- Group with remote monitoring: All patients seen in hospital and for whom the doctor will choose whether or not to offer one of the 2 solutions, alone or in combination, will be considered as included in the study, and their non-objection will be collected.
  Subsequently, patients will benefit from follow-up for 6 months: V0 inclusion visit- V1 telephone contact at 1 month optional only for patients participating in one of the 2 programs and V2 consultation at 6 months. The 0 and 6M visits are part of the usual follow-up of patients hospitalized for heart failure.
  Administration of questionnaires:
  * Girerd's questionnaire on therapeutic compliance
  * SUTAQ inspired digital tools acceptability questionnaire: only for patients with remote monitoring
  * SSQ6 social support questionnaire
  Interventions: Device: Remote monitoring
- Group without intervention: All patients seen in hospital and for whom the doctor will choose whether or not to offer one of the 2 solutions, alone or in combination, will be considered as included in the study, and their non-objection will be collected.
  Subsequently, patients will benefit from follow-up for 6 months: V0 inclusion visit- V1 telephone contact at 1 month optional only for patients participating in one of the 2 programs and V2 consultation at 6 months. The 0 and 6M visits are part of the usual follow-up of patients hospitalized for heart failure.
  Administration of questionnaires:
  * Girerd's questionnaire on therapeutic compliance
  * SSQ6 social support questionnaire

INTERVENTIONS:
Other: PRADO-IC — The CAM (Health Insurance Advisor) are part of the staff of the Primary Health Insurance Funds (CPAM). They are physically present in the establishments participating in the PRADO.
  They are facilitators between city health professionals and the patient for their return home.
  They assist the patient in making appointments with their general practitioner, their cardiologist, and the IDE (general care nurses) trained at PRADO-IC who will make the home visits.
  After returning home, the CAM verifies, by two telephone calls at 1 week and 2 months, that the patient has initiated his outpatient follow-up.
  IDE, trained in the therapeutic education of the IC patient according to the PRADO-IC device, carry out:
  * for NYHA (New York Heart Association) 1-2 patients: 8 home visits in two months.
  * for NYHA 3-4 patients: 8 home visits in 2 months, upon confirmation and prescription from the physician, 8 visits in the following 4 months.
  The doctor carries out a long consultation at 2 months.
  Groups: Group with PRADO; Group with PRADO + remote monitoring
Device: Remote monitoring — Chronic Care Connect is intended for remote medical monitoring of patients suffering from chronic heart failure.
  It consists of a web application (named NOMHADChronic™) and non-medical remote human assistance performed by qualified personnel.
  Non-medical human assistance allows the following steps to be carried out:
  * characterization of alerts
  * structured follow-up of remote patients.
  This non-medical human assistance is provided by:
  * nurses trained in therapeutic education and cardiology, Customer Relations Advisors, and logisticians.
  Weight and symptoms (listed in an 8-question questionnaire) are collected respectively using a connected scale and the mobile application.
  It allows, via a web browser:
  * to the personnel constituting the non-medical human assistance, to have access to the health data of the patients
  * remote monitoring doctors, to have access to the health data of each of their own patients, and to carry out medical remote monitoring procedures.
  Groups: Group with PRADO + remote monitoring; Group with remote monitoring

SUMMARY:
Patients with heart failure (HF), after hospitalization, present a marked fragility. Interventions improving the coordination of care actors at the time of discharge from hospitalization have been tested and have shown, in preliminary studies, a reduction in rehospitalizations for heart failure and all-cause mortality.

Among these promising devices, two have recently been deployed nationwide.

* The return home program for IC patients (PRADO IC), set up by the Health Insurance, aims to facilitate the return and stay at home after hospitalization. It offers assistance with the initiation of outpatient medical follow-up, nursing follow-up for 2 to 6 months depending on the severity of the patient, and a follow-up log facilitating the exchange of information.
* At the same time, as part of the ETAPES (Telemedicine experiments for the improvement of healthcare pathways) program of the Health Insurance, the deployment of telemedicine for remote monitoring of heart failure pursues a comparable objective of reducing rehospitalizations.

These two systems are widely deployed on a national scale, and are intended to be universal.

Our hypothesis is that adherence to care transition and telemedicine programs, and therefore their effectiveness, may depend on their association, as well as socio-demographic, cultural, and geographical factors.

DETAILED DESCRIPTION:
Patients with heart failure (HF), after hospitalization, present a marked fragility: in France, in the first year, 29% die and 45% are rehospitalized for HF. Interventions improving the coordination of care actors at the time of discharge from hospitalization have been tested and have shown in preliminary studies a reduction in rehospitalizations for HF (relative risk (RR) from 0.51 to 0.74) and all-cause mortality (RR 0.75 to 0.87).

Among these promising devices, two have recently been deployed nationwide.

* The return home program for IC patients (PRADO IC), set up by the Health Insurance, aims to facilitate the return and stay at home after hospitalization. It offers assistance with the initiation of outpatient medical follow-up, nursing follow-up for 2 to 6 months depending on the severity of the patient, and a follow-up log facilitating the exchange of information. It is based on the assumption that these actions will improve the coordination of care between the hospital and the city, and between home nurses and doctors. In addition, nurses reinforce therapeutic patient education (TPE), whether or not it is initiated in a setting dedicated to TPE.
* At the same time, as part of the ETAPES program of the Health Insurance, the deployment of telemedicine for remote monitoring of heart failure pursues a comparable objective of reducing rehospitalizations. It is based on the hypothesis that the early signs of cardiac decompensation can be diagnosed by telemonitoring and trigger earlier and therefore less aggressive management for similar effectiveness.

These two systems are widely deployed on a national scale, and are intended to be universal.

However, three points can call into question the effectiveness of this deployment: their evaluation is often difficult, the extrapolability of randomized studies to health systems and different populations is low, and the complementarity of two independently constructed programs has never been been studied so far.

1. The preliminary data concerning the PRADO were epidemiological, historical, comparative before-elsewhere, on the SNIIRAM (National health insurance inter-scheme information system) databases, without optimal consideration of clinical and cultural confounding factors.
2. The acceptability of these programs by all health professionals (and therefore how they choose to deploy such and such a system for a given patient) and patients in the French context is not known.
3. The PRADO system and telemedicine solutions, acting differently, could be synergistic and therefore multiply the benefits obtained. However, in practice, some patients experience these programs as intrusive, and it is possible that their adherence is in fact all the worse when two programs are implemented. Similarly, from the prescriber's point of view, the way in which the various possible combinations are chosen is unknown.

The answer to these three questions is necessary to guide the most effective deployment of these programs nationwide.

Our hypothesis is that adherence to care transition and telemedicine programs, and therefore their effectiveness, may depend on their association, as well as socio-demographic, cultural, and geographical factors.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient hospitalized at the time of inclusion for cardiac decompensation, or cause of admission for which heart failure plays a decisive or aggravating role (co-infection, etc.) recognized by the clinician.
* Patient agreeing to take part in this research (absence of non-objection)

Exclusion Criteria:

* Refusal to participate
* Pregnant or breastfeeding women, patients unable to give protected adult consent, vulnerable people (art.L.1121-6, L.1121-7, L.1211-8, L.1211-9)
* Subject deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population consists of adult patients, suffering from heart failure, hospitalized for cardiac decompensation.
  The source population consists of patients hospitalized for heart failure in cardiology departments of UH of Montpellier, Nîmes, Bassin de Thau and Béziers.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients participating in heart failure programs at 1 month | At 1 month
  Participation corresponds to:
  * for the PRADO group: visits to the attending physician and home nurses, and appointments made with the cardiologist
  * for the remote monitoring group: completion of at least 80% of the weighings
Percentage of patients participating in heart failure programs at 6 months | At 6 months
  Participation corresponds to:
  * for the PRADO group: visits to the attending physician and home nurses, and appointments made with the cardiologist
  * for the remote monitoring group: completion of at least 80% of the weighings
  * for the group without intervention: completion of the visit at 6 months

SECONDARY OUTCOMES:
Number of non-participation of patients | At inclusion
  Describe the causes of non-participation, primary (when the intervention was proposed)
Number of non-participation of patients | through study completion, an average of 6 months
  Describe the causes of non-participation secondary (after initial acceptance)
Percentage effectiveness of pathology programs at 1 month | between inclusion and 1 month
  Evaluate the effectiveness at 1 month of the PRADO and telemedicine programs, as well as their interaction, on hospitalizations for all causes combined
Percentage effectiveness of pathology programs at 1 month | between inclusion and 1 month
  Evaluate the effectiveness at 1 month of the PRADO and telemedicine programs, as well as their interaction, on hospitalizations for heart failure
Percentage effectiveness of pathology programs at 1 month | between inclusion and 1 month
  Evaluate the effectiveness at 1 month of the PRADO and telemedicine programs, as well as their interaction, on deaths from all causes combined
Percentage effectiveness of pathology programs at 1 month | between inclusion and 1 month
  Evaluate the effectiveness at 1 month of the PRADO and telemedicine programs, as well as their interaction, on deaths due to heart failure
Percentage effectiveness of pathology programs at 6 months | between inclusion and 6 months
  Evaluate the effectiveness at 1 month of the PRADO and telemedicine programs, as well as their interaction, on hospitalizations for all causes combined
Percentage effectiveness of pathology programs at 6 months | between inclusion and 6 months
  Evaluate the effectiveness at 1 month of the PRADO and telemedicine programs, as well as their interaction, on hospitalizations for heart failure
Percentage effectiveness of pathology programs at 6 months | between inclusion and 6 months
  Evaluate the effectiveness at 1 month of the PRADO and telemedicine programs, as well as their interaction, on deaths from all causes combined
Percentage effectiveness of pathology programs at 6 months | between inclusion and 6 months
  Evaluate the effectiveness at 1 month of the PRADO and telemedicine programs, as well as their interaction, on deaths due to heart failure
percentage of effectiveness on the course of care at 6 months | between inclusion and 6 months
  Average number of consultations per month with the general practitioner
percentage of effectiveness on the course of care at 6 months | between inclusion and 6 months
  Time between the first consultation with the general practitioner and discharge from hospital
percentage of effectiveness on the course of care at 6 months | between inclusion and 6 months
  Average number of consultations per month with the cardiologist
percentage of effectiveness on the course of care at 6 months | between inclusion and 6 months
  Time between the first consultation with the cardiologist and discharge from hospital
percentage of days with at least one nursing contact | between inclusion and 6 months
  number of days with at least one nursing contact
Number of emergency medical contacts | between inclusion and 6 months
  are considered as emergency contacts: consultations with emergency increase, or increase for Night, Weekend or Public Holiday; consultations in emergencies; hospitalizations with emergency entry mode
percentage of medical appointments made | between inclusion and 6 months
  according to the continuity of care index, corresponding to the percentage of appointments made by patients with a doctor
Average number of treatment days taken per patient per month | between inclusion and 6 months
  For taking sartans treatments
Average number of treatment days taken per patient per month | between inclusion and 6 months
  For taking beta-blocker treatments
Average number of treatment days taken per patient per month | between inclusion and 6 months
  Coefficient of variation of the daily dose of loop diuretics, calculated as the average dose between two deliveries
percentage of efficiency on the cost of the care pathway at 6 months | between inclusion and 6 months
  Cost of care pathways: made up of production costs over 6 months after initial hospitalization, and includes all direct costs, whether medical or non-medical.
percentage of physicians offering heart failure programs | between inclusion and 6 months
  Beliefs of physicians on the facilitating elements and on the obstacles of these programs

CONTACTS AND LOCATIONS:
Overall Officials: François ROUBILLE, PUPH, Principal Investigator — UH of Montpellier
Locations (1):
- University Hospital, Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided